CLINICAL TRIAL: NCT06712303
Title: Role of Multi-detector CT and MRI in Diagnosis of Congenital Inner Ear Anomalies
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Khaled Fahmi, Principal Investigator, Assiut University
Other Study IDs: CT,MRI in inner ear anomalies
Record Dates: First submitted 2024-11-22; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Ear Disease, Inner
Keywords: MRI; Ct; Ear disease
MeSH Terms: conditions — Labyrinth Diseases; Ear Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: MRI ,ct — Every patient will be subjected to
  1. MSCT examination: All patients will undergo MSCT (Siemens somatom 32 slice ,16 slice ,GE bright speed 16 slice ) Non contrast high-resolution CT of the temporal bone with the following parameters:{ 0.75-mm collimation, 130 kvp, 20 mA, topogram length 265}. Patients will be scanned in the supine position with craniocaudal direction. Scanning will be parallel to the orbito-meatal line from the lower margin of the external auditory meatus and extended upward to the arcuate eminence of the superior semicircular canal, as seen on the lateral topogram. Followed by image reconstruction in both the axial and coronal planes to evaluate the inner ear and its malformations, The initial data sets will be reconstructed at 0.6 mm slice thickness. The raw axial image data set can be reconstructed with a section thickness of as little as 0.3 mm to obtain high-quality coronal reformatted images. A 512 × 512 matrix is used, and all the images are reviewed wit

SUMMARY:
Evaluation of combined value of Multi-detector computed tomography (MDCT) and Magnetic resonance imaging (MRI) in the diagnosis of congenital abnormalities of the inner ear and internal auditory canal in patients with congenital hearing loss and preoperative evaluation of cochlear implant candidates.

DETAILED DESCRIPTION:
Introduction:

Inner ear malformation (IEM) with associated sensoryneural hearing loss (SNHL) is a major cause of childhood disability.

The embryology of the inner ear must be known as many of the inner ear malformations present as a result of the arrest during the various stages of embryology.

Congenital malformations of the inner ear may be considered in two broad categories:

1. malformations with pathologic changes that involve only the membranous labyrinth.
2. malformations that involve both the osseous and the membranous labyrinth.

Congenital sensorineural hearing loss arises as a result of abnormalities in the inner ear, the vestibulocochlear nerve, or the processing centres of the brain. The abnormality may have a genetic cause or be a sequel of infection or injury at birth; in some cases, no cause is identified.

One of the paths in the investigation of congenital sensorineural hearing loss (CSNHL) is to try to characterize its aetiology through the inner ear evaluation using high resolution computer tomography (CT) scans. With minor malformation, it is not always possible for a simple visual inspection to recognize if the structure in the inner ear is normal or not.

Both CT and MR can be used to look at inner ear malformations but often both techniques are complementary. CT is preferred when associated middle or external ear malformations must be excluded. Magnetic resonance is preferred when subtle changes in the membranous labyrinth or abnormalities of the nerves in the internal auditory canal must be visualised Moreover, some changes inside the membranous labyrinth can only be seen on sub-millimetric heavily T2-weighted MR images.

Only MR can demonstrate the abnormal course, hypoplasia or aplasia of the vestibulocochlear nerve (or one of is three branches) and facial nerve.

HRCT and MRI temporal bone are complementary to each other in evaluating children for cochlear implantation as HRCT is excellent for demonstrating bony details but, lack in providing details of inner ear neural structures and MRI is better than CT in demonstrating vestibulocochlear nerves.

Combined HRCT and MRI studies are mandatory for evaluation of inner ear, the radiologist must be familiar with imaging findings that absolutely contraindicate implantation (Cochlear aplasia, cochlear nerve aplasia and labyrinthine aplasia), and with those that relatively contraindicate implantation (labyrinthitis ossificans, other inner ear dysplasia) and with other findings that could significantly alter or complicate surgery (hypo plastic mastoid process, facial nerve dehiscence, oto-mastoiditis)

ELIGIBILITY:
Inclusion Criteria:

* all patient of inner ear anomalies

Exclusion Criteria:

* studied groups ,mri

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any age group come for cochlear implantation
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Inner ear anomalies detection by CT and MRI | Baseline
  accurate and early diagnosis of patsuffer from suffer from sensory neural hearing loss (SNHL)

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Y. Mohamed, Study Director — Assistant professor doctor; Hossam E. Mohamed, Study Director — Professor doctor

IPD SHARING:
Plan to Share IPD: No